CLINICAL TRIAL: NCT02502656
Title: RAS Mutation Testing in the Circulating Blood of Patients With Metastatic Colorectal Cancer: Concordance With the "Standard" Testing Method From Tumor Tissue and Review of Associated Timelines and Costs
Brief Title: RAS Mutation Testing in the Circulating Blood of Patients With Metastatic Colorectal Cancer
Acronym: RASANC
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Association des Gastroentérologues Oncologues (Other)
Responsible Party: Sponsor
Other Study IDs: RASANC
Record Dates: First submitted 2015-07-16; First posted 2015-07-20 (Estimated); Last update posted 2016-11-17 (Estimated); Status verified 2016-11

CONDITIONS: Colorectal Cancer
Keywords: RAS mutation; DNA; Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood collection will be performed on the day of the first oncological consultation
Oversight: Data Monitoring Committee: No

SUMMARY:
This study will evaluate the concordance of RAS mutation detection between the results obtained from circulating tumor DNA and those obtained with the "standard" method (testing from tumor tissue).

ELIGIBILITY:
Inclusion Criteria:

* Pathologically confirmed metachronous or synchronous metastatic colorectal cancer
* No prior chemotherapy with the exception of adjuvant chemotherapy completed ≥ 6 months prior to enrollment
* Signed written informed consent obtained prior to any study specific screening procedures
* Patients willing to provide a blood sample for Translational Research

Exclusion Criteria:

* No tumor block available
* Previous malignancy in the last 5 years
* Medical, sociological, psychological or legal conditions that would not permit the patient to sign informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All treatment naive patients seen in consultation for metastatic colorectal cancer in the participating centers
Sampling Method: Non-Probability Sample
Enrollment: 425 (Estimated)
Dates: Start 2015-07; Primary Completion 2017-08 (Estimated); Study Completion 2017-08 (Estimated)

PRIMARY OUTCOMES:
Concordance regarding the mutation of RAS (yes vs no, dichotomous variable) between the two methods | Baseline
  RAS mutations will be compared between tumor tissue (standard testing methods) and results obtained from circulating tumor DNA

SECONDARY OUTCOMES:
Concordance regarding the mutation of RAS (yes vs no, dichotomous variable) between the two methods in patients for whom circulating tumor DNA has been identified in the avalaible plasma sample. | Baseline
  RAS mutations will be compared between tumor tissue (standard testing methods) and results obtained from circulating tumor DNA. This subgroup of patients is defined as patients with at least one mutation identified in the panel of tested genes (Ion AmpliSeq Colon and Lung Cancer Panel) (RAS mutation or mutations on other genes TP53, PIK3CA, SMAD4 .... ) or with at least one methylated biomarker identified (for patients with no mutation identified in the panel of genes tested).
Comparison of the timelines to obtain results between the two methods | Baseline
  Timelines to obtain RAS mutations will be compared between tumor tissue (standard testing methods) and circulating tumor DNA
Comparisons of the costs between the two methods | Baseline
  Costs for the two methods will be compared between tumor tissue (standard testing methods) and circulating tumor DNA

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Baptiste Bachet, Dr, Principal Investigator — Association des Gastro-entérologues Oncologues (AGEO)
Locations (14):
- France (14):
  - Hôpital Avicenne, Bobigny
  - Hopital Béclère, Clamart
  - Hopital Henri Mondor, Créteil
  - Hopital Kremlin-Bicêtre, Le Kremlin-Bicêtre
  - CH Longjumeau et Sud, Longjumeau
  - Hopital Mermoz, Lyon
  - Hopital Cochin, Paris
  - Hopital Saint-Antoine, Paris
  - Hopital Saint-Louis, Paris
  - Hôpital Européen Georges Pompidou, Paris
  - Hôpital Pitié Salpêtrière, Paris
  - CHU Poitiers, Poitiers
  - CHU Robert Debré, Reims
  - Hôpital Trousseau, Tours

REFERENCES:
- [Derived] Bachet JB, Laurent-Puig P, Meurisse A, Bouche O, Mas L, Taly V, Cohen R, Gornet JM, Artru P, Louafi S, Thirot-Bidault A, Baumgaertner I, Coriat R, Tougeron D, Lecomte T, Mary F, Aparicio T, Marthey L, Blons H, Vernerey D, Taieb J. Circulating tumour DNA at baseline for individualised prognostication in patients with chemotherapy-naive metastatic colorectal cancer. An AGEO prospective study. Eur J Cancer. 2023 Aug;189:112934. doi: 10.1016/j.ejca.2023.05.022. Epub 2023 Jun 7. PMID 37390800
- [Derived] Bachet JB, Bouche O, Taieb J, Dubreuil O, Garcia ML, Meurisse A, Normand C, Gornet JM, Artru P, Louafi S, Bonnetain F, Thirot-Bidault A, Baumgaertner I, Coriat R, Tougeron D, Lecomte T, Mary F, Aparicio T, Marthey L, Taly V, Blons H, Vernerey D, Laurent-Puig P. RAS mutation analysis in circulating tumor DNA from patients with metastatic colorectal cancer: the AGEO RASANC prospective multicenter study. Ann Oncol. 2018 May 1;29(5):1211-1219. doi: 10.1093/annonc/mdy061. PMID 29438522